CLINICAL TRIAL: NCT04484493
Title: Role of Corticosteroid Nasal Spray in Recovery of Smell Sensation in COVID-19 Patients
Brief Title: Corticosteroid Nasal Spray in COVID-19 Anosmia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Abdelalim, MD lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 4-7-2020
Record Dates: First submitted 2020-07-22; First posted 2020-07-23 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Anosmia
Keywords: covid19; anosmia; mometasone nasal spray
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mometasone nasal spray (Experimental): Patients will receive topical corticosteroid nasal spray (mometasone furoate nasal spray) in appropriate dose of 2 puff in each nostril (100 µg once daily) beside olfactory training.
  Interventions: Drug: mometasone furoate nasal spray
- control (No Intervention): Patients will not receive topical corticosteroid nasal spray but only olfactory training.

INTERVENTIONS:
Drug: mometasone furoate nasal spray — dose of 2 puff in each nostril (100 µg once daily each nostril).
  Other Names: steroid nasal spray
  Arms: mometasone nasal spray

SUMMARY:
The aim of this study is to evaluate the role of the topical corticosteroids nasal spray (mometasone furoate nasal spray) in improving anosmia in patients recovered from COVID-19 infection.

DETAILED DESCRIPTION:
This study willbe submitted on patients who recently recovered from proven COVID-19 infection and complaining of anosmia or hyposmia.The proven COVID-19 infection will be relied on a positive real-time reverse transcription polymerase chain reaction (rRT-PCR) with samples obtained by a nasopharyngeal swab. The recovery is defined as 2 consecutives negative (rRT-PCR) samples.

Complete medical history will be taken, and essential clinical assessment with appropriate protective measures will be performed in all patients.The patients in the study will be randomly divided into two groups: - Group I: -who will receive topical corticosteroid nasal spray (mometasone furoate nasal spray) beside olfactory training Group II: -who will not receive topical corticosteroid nasal spray but only olfactory training.

As regards the assessment of smell,the patient will assess his smell sensation using familiar substances with distinctive odor. A jar of coffee, a branch of mint and garlic are some used substances. The patient will report the degree of anosmia subjectively with score on a scale from 0 to 10.The assessment of smell will be done initially after recovery/discharge, after 1 week, 2 weeks and after 3 weeks for all patients. The duration of smell loss will be recorded from the onset of anosmia till full recovery of the sensation.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 yrs or older patients
* confirmed case (+ve PCR),
* recovered/discharged (2 -ve PCR),
* suffered from sudden recent anosmia or hyposmia

Exclusion Criteria:

* patients already on nasal steroid
* with previous chronic rhinological pathologies,
* patients on systemic steroid for previous systemic disease,
* anosmia improved before COVID19 recovery,
* pregnancy
* patients who will not complete the follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
improvement of olfaction | 3 weeks
  The patient will report the degree of anosmia subjectively with score on a scale from 0 to 10 (0 means total loss of smell and 10 refers to completely normal smell sensation).

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman A Abdelalim, MD, Principal Investigator — Benha University; Rasha A Elsayed, MD, Study Chair — Benha University; Mona A Elawady, MD, Study Chair — Benha University; Abdelhakim F Ghallab, MD, Study Chair — Benha University; Ayman A Mohamady, MD, Study Chair — Benha University
Locations (1):
- Benha University Hospital, Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heilmann S, Just T, Goktas O, Hauswald B, Huttenbrink KB, Hummel T. [Effects of systemic or topical administration of corticosteroids and vitamin B in patients with olfactory loss]. Laryngorhinootologie. 2004 Nov;83(11):729-34. doi: 10.1055/s-2004-825676. German. PMID 15538662
- [Background] Hura N, Xie DX, Choby GW, Schlosser RJ, Orlov CP, Seal SM, Rowan NR. Treatment of post-viral olfactory dysfunction: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2020 Sep;10(9):1065-1086. doi: 10.1002/alr.22624. Epub 2020 Jun 25. PMID 32567798
- [Derived] Webster KE, O'Byrne L, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the prevention of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013877. doi: 10.1002/14651858.CD013877.pub3. PMID 36063364
- [Derived] Abdelalim AA, Mohamady AA, Elsayed RA, Elawady MA, Ghallab AF. Corticosteroid nasal spray for recovery of smell sensation in COVID-19 patients: A randomized controlled trial. Am J Otolaryngol. 2021 Mar-Apr;42(2):102884. doi: 10.1016/j.amjoto.2020.102884. Epub 2021 Jan 4. PMID 33429174